CLINICAL TRIAL: NCT01908959
Title: Madres Para la Salud (Mothers for Health)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Colleen Keller, Colleen Keller, PhD, RN-C, FNP, FAHA, FNAP, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1R01NR010356-01A2 (NIH)
Record Dates: First submitted 2013-07-19; First posted 2013-07-26 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Overweight and Obesity; Depression, Postpartum; Mother (Person)
Keywords: Hispanic Women; Postpartum; Overweight Hispanic Women; Low-income; Physical Activity; Walking
MeSH Terms: conditions — Overweight; Obesity; Depression, Postpartum; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Madres para la Salud (Experimental): Participants attended Madres para la Salud sessions in a group, led by a promotora at the Maricopa Medical Center and other community based sites. Sessions consisted of a 30 minute education and social support session where women learned to walk at least 150 minutes a week at a 20 minute-mile pace, and up to 30 minutes of moderate intensity walking with the group. Participants received an Omron pedometer and learned to monitor walking intensity. Participants set and reviewed weekly walking goals at the group sessions and recorded aerobic steps per day. After the 12 week sessions, participants met with the promotora once a week for 40 weeks, in-group, to walk at a moderate intensity for 30 minutes, to download and review pedometer data. Data was collected at baseline, 3, 6, 9 and 12 months.
  Interventions: Behavioral: Madres para la Salud
- Attention-control (No Intervention): Participants in the attention receive monthly brief telephone calls by research technicians and collection of study data on-site at the Maricopa Medical Center and other community based sites at baseline, 6, and 12 months (T1, T3, T5). The staff did not give advice or support specific to walking, which enabled a valid evaluation of the intervention effect. The content given to the attention-control group did not include the "active ingredients" of the Madres para la Salud intervention. The attention-control group received monthly mailings of health-related information regarding common postpartum or newborn concerns, such as breastfeeding, infant sleep, sibling rivalry, emotional support related to new parenthood, and early childhood development topics.

INTERVENTIONS:
Behavioral: Madres para la Salud — Participants attended Madres para la Salud sessions in a group, led by a promotora at the Maricopa Medical Center and other community based sites. Sessions consisted of a 30 minute education and social support session where women learned to walk at least 150 minutes a week at a 20 minute-mile pace, and up to 30 minutes of moderate intensity walking with the group. Participants received a pedometer and learned to monitor their walking intensity. Participants set and reviewed weekly walking goals at the group sessions and recorded aerobic steps per day. After the 12 week sessions, participants met with the promotora once a week for 40 weeks of in-group walking at a moderate intensity for 30 minutes, to download and review pedometer data. Data was collected at baseline, 3, 6, 9 and 12 months.
  Arms: Madres para la Salud

SUMMARY:
The purpose of "Madres Para la Salud" [Mothers for Their Health] is to see how support and encouragement can help women to make positive changes in their health. This program tested if supportive information, encouragement, and walking as a group would increase physical activity and health benefits, such as weight loss and postpartum depression.

Participants in this study were randomly assigned to one of two groups, a walking or a non-walking group. The walking group met weekly. Participants were given a pedometer to record the number of steps taken daily.

Participants met one time each week with our study staff. Participants walked four other days per week on their own, or with other group members. Participants measurements included body fat, waist, and hip at the beginning of the study, and at 3, 6, 9, and 12 months. The non-walking group received a weekly mailed newsletter about topics such as parenting, infant growth and development, and reproductive health. Non-walking group participants' measurements included body fat, waist, and hip at the beginning of the study and at 6 and 12 months.

DETAILED DESCRIPTION:
Project Summary

The purpose of "Madres para la Salud" (Mothers for Health) was to explore the effectiveness of a culturally specific intervention using walking "bouts" to affect changes in the health of Hispanic women following childbirth. The project will advance our understanding of the relationship between moderate increases in physical activity and consequent body fat loss and decreased postpartum depression symptoms in sedentary Hispanic women during the postpartum period. This was accomplished by having a group of women who participated in supportive information and walking sessions, both alone and with study personnel, and an attention control group who received monthly phone calls to address common postpartum health concerns, but who did not participate in the walking program. Both groups received weekly health-focused newsletters with no content related to the intervention. The women had a random assignment to a group.

Study Aims

The purpose of this social support intervention program was to test the theory-driven Madres para la Salud with Hispanic women by conducting a formative evaluation of the intervention:

Aim 1: Examine the effectiveness of the Madres para la Salud, a theoretically driven social support intervention for reducing the distal outcomes in: (a) body fat; (b) systemic and fat tissue inflammation; and (c) PPD symptoms among postpartum Hispanic women compared with an attention control group, at 6 and 12 months, after controlling for dietary intake.

Aim2: Test whether the theoretical mediators, intermediate outcomes, of social support and walking, and environmental factor moderators, affect changes in body fat; systemic and fat tissue inflammation; and PPD symptoms among postpartum Hispanic women completing the Madres para la Salud intervention compared with an attention control group, at 6 and 12 months, after controlling for dietary intake.

Aim 3: Determine the relationship between the immediate outcome of walking (minutes walked per week) and change in the distal outcomes of: (a) body fat; (b) systemic and fat tissue inflammation; and (c) PPD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic descendent
* Between 18 and 40 years old
* At least 6-weeks but less than 6-months post childbirth
* Sedentary (according to the American College of Sports Medicine)
* Have the ability to participate in moderate intensity physical activity (according to the Physical Activity Readiness Questionnaire (PAR-Q))

Exclusion Criteria:

* Pregnant or planning a pregnancy in the next 12 months
* Have a BMI less than 25 or greater than 35
* Take anti-depressant medications
* Take anticoagulants or herbal therapy to thin the blood
* Participate in regular, strenuous physical activity (exceeding 150 minutes of moderate physical activity per week)
* Severe musculoskeletal or cardiorespiratory problems that would preclude physical activity
* Infectious illness
* Acute inflammation (white blood count outside the normal range of 4.8-10.8 of 1000/mm3)
* Chronic systemic inflammatory diseases (e.g., rheumatoid arthritis), or other acute illness that may affect systemic inflammation at the time of blood draw and fat tissue biopsy
* Regularly taking high doses of oral steroid medication (more than typical basal replacement levels)
* High doses of aspirin (above 1 g/day), or high doses of nonsteroidal anti-inflammatory drugs (e.g., 3-4 times/day)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 177 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Body Fat Percentage at 6 months | 6 months
  Body fat was measured using bioelectric impedance (BIA), with portable four-terminal BIA measurement system (Tanita Corporation of America, Inc, Arlington Heights, IL). Instrument calibration was performed internally prior to each estimate of body composition. Measurement of body composition using BIA analysis followed the method outlined by Ritchie, Miller, and Smiciklas-Wright (Ritchie, Miller, & Smiciklas-Wright, 2005). A subsample of the intervention group had body fat measured with state-of-the-art dual energy x-ray absorptiometry (DEXA) at baseline and 12 months.
Change from Baseline Body Fat Percentage at 12 months | 12 Months
  Body fat was measured using bioelectric impedance (BIA), with portable four-terminal BIA measurement system (Tanita Corporation of America, Inc, Arlington Heights, IL).
Change from Baseline Systemic and fat tissue inflammation at 12 months | 12 months
  Systemic and fat tissue inflammation was measured through a fat biopsy that was conducted by a trained physician (M.D.)
Change from Baseline in Edinburgh Postnatal Depression Scale at 6 months | 6 months
  Postpartum Depression Symptoms were measured with the Edinburgh Postnatal Depression Scale (EPDS)questionnaire.
Change from Baseline in Edinburgh Postnatal Depression Scale at 12 months | 12 months
  Postpartum Depression Symptoms were measured with the Edinburgh Postnatal Depression Scale (EPDS)questionnaire.

SECONDARY OUTCOMES:
Change from baseline in Medical Outcomes Study (MOS) Social Support Survey at 6 months | 6 months
  Social Support and walking were measured through the MOS Social Support survey and the Social Support and Exercise Survey.
Change from baseline in Medical Outcomes Study (MOS) Social Support Survey at 12 months | 12 months
  Social Support was measured through the MOS Social Support survey and the Social Support and Exercise Survey.
Change from baseline in Neighborhood Health Questionnaire at 6 months | 6 months
  Environmental Factor Moderators were measured through the Neighborhood Health Questionnaire. This questionnaire includes questions relating to Neighborhood walkability, Aesthetic Quality, Safety, Social Cohesion, Violence, and Activities with neighbors.
Change from baseline in Neighborhood Health Questionnaire at 12 months | 12 months
  Environmental Factor Moderators were measured through the Neighborhood Health Questionnaire. This questionnaire includes questions relating to Neighborhood walkability, Aesthetic Quality, Safety, Social Cohesion, Violence, and Activities with neighbors.

OTHER OUTCOMES:
Relationship between Walking Outcomes and listed Primary Outcomes at 6 months | 6 months
  The relationship between walking outcomes and the previously listed primary outcomes was measured through the change in body fat and postpartum depression symptoms (at Baseline, 6 months, and 12 months), systemic and fat tissue inflammation (at Baseline and 12 months).
Relationship between Walking Outcomes and listed Primary Outcomes at 12 months | 12 months
  The relationship between walking outcomes and the previously listed primary outcomes was measured through the change in body fat and postpartum depression symptoms (at Baseline, 6 months, and 12 months), systemic and fat tissue inflammation (at Baseline and 12 months).

CONTACTS AND LOCATIONS:
Overall Officials: Colleen S Keller, PhD, Principal Investigator — Arizona State University, College of Nursing and Health Innovation
Locations (1):
- Maricopa Integrated Health System, Phoenix, Arizona, United States

REFERENCES:
- [Background] Records K, Keller C, Ainsworth B, Permana P. Instrument selection for randomized controlled trials: why this and not that? Contemp Clin Trials. 2012 Jan;33(1):143-50. doi: 10.1016/j.cct.2011.09.006. Epub 2011 Oct 1. PMID 21986392
- [Background] Keller C, Records K, Ainsworth B, Belyea M, Permana P, Coonrod D, Vega-Lopez S, Nagle-Williams A. Madres para la Salud: design of a theory-based intervention for postpartum Latinas. Contemp Clin Trials. 2011 May;32(3):418-27. doi: 10.1016/j.cct.2011.01.003. Epub 2011 Jan 14. PMID 21238614
- [Background] Keller C, Todd M, Ainsworth B, Records K, Vega-Lopez S, Permana P, Coonrod D, Nagle Williams A. Overweight, obesity, and neighborhood characteristics among postpartum Latinas. J Obes. 2013;2013:916468. doi: 10.1155/2013/916468. Epub 2013 Feb 6. PMID 23476752
- [Background] Ainsworth BE, Keller C, Herrmann S, Belyea M, Records K, Nagle-Williams A, Vega-Lopez S, Permana P, Coonrod DV. Physical activity and sedentary behaviors in postpartum Latinas: Madres para la Salud. Med Sci Sports Exerc. 2013 Jul;45(7):1298-306. doi: 10.1249/MSS.0b013e3182863de5. PMID 23439416
- [Derived] Vega-Lopez S, Pignotti GA, Keller C, Todd M, Ainsworth B, Nagle Williams A, Records K, Coonrod D, Permana P. Participation in a Social-Support Physical Activity Intervention Modestly Improves Lipoprotein Cholesterol Distribution Among Postpartum Sedentary Hispanic Women. J Phys Act Health. 2015 Sep;12(9):1289-97. doi: 10.1123/jpah.2014-0245. Epub 2014 Nov 19. PMID 25408998
- [Derived] Keller C, Ainsworth B, Records K, Todd M, Belyea M, Vega-Lopez S, Permana P, Coonrod D, Nagle-Williams A. A comparison of a social support physical activity intervention in weight management among post-partum Latinas. BMC Public Health. 2014 Sep 19;14:971. doi: 10.1186/1471-2458-14-971. PMID 25233867